CLINICAL TRIAL: NCT05462938
Title: Comparative Study of Propofol Versus Dexmedetomidine for Conscious Sedation During Transcatheter Aortic Valve Implantation
Brief Title: Conscious Sedation for Transcatheter Aortic Valve Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Agathi Karakosta, Assistant Professor of Anaesthesiology, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11772
Record Dates: First submitted 2022-07-08; First posted 2022-07-18 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Renal Function Disorder; Postoperative Delirium; Adverse Event; Death; Satisfaction
Keywords: transcatheter aortic valve replacement; dexmedetomidine; propofol; conscious sedation; monitored anesthesia care
MeSH Terms: conditions — Emergence Delirium; Death; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol group (Active Comparator): Continuous infusion of propofol
  Interventions: Drug: Continuous infusion of propofol
- Dexmedetomidine group (Active Comparator): Continuous infusion of dexmedetomidine
  Interventions: Drug: Continuous infusion of dexmedetomidine

INTERVENTIONS:
Drug: Continuous infusion of propofol — Sedation under continuous infusion of propofol. Small doses of fentanyl will be administered if needed.
  Other Names: Prop Group
  Arms: Propofol group
Drug: Continuous infusion of dexmedetomidine — Sedation under continuous infusion of dexmedetomidine. Small doses of fentanyl will be administered if needed.
  Other Names: Dex Group
  Arms: Dexmedetomidine group

SUMMARY:
Aortic valve stenosis is the heart valve disease with the highest prevalence among the elderly, and may lead to heart failure. Until recently, the only definitive treatment was surgical replacement (SAVR). However, the increased risk associated with the surgical procedure excluded patients with multiple co-morbidities. As the population is aging and more and more patients may present with aortic stenosis, the need of a less invasive approach has emerged. Transcatheter Aortic Valve Replacement (TAVR) offered an alternative therapy for these high risk patients. This new method has seen worldwide acceptance, has been proven very beneficial for these patients, and therefore its indications have been expanded to intermediate risk patients, as well. Until recently, general anesthesia was the primary anesthetic technique for TAVR, but conscious sedation or monitored anesthesia care (MAC) is gaining more and more popularity lately. Our knowledge regarding the comparison between general anesthesia and MAC in TAVR procedures is derived mainly from observational studies and few randomized trials. MAC seems to be associated with less inotropic drug usage, shorter procedural times, shorter intensive care unit (ICU) and hospital length of stay. However, according to published data, there were no differences in 30-day mortality and complications between these two techniques.

Even less are known about the most suitable anesthetic agent for MAC during TAVR. Many drugs have been used, with propofol and dexmedetomidine being the most popular. However, there are only few comparative studies and their results are not conclusive.

This study compares MAC under propofol and MAC under dexmedetomidine for TAVR in order to examine which method of conscious sedation comes with more beneficial postoperative outcomes for the patients.

DETAILED DESCRIPTION:
Aortic valve stenosis is the most common heart valve disease among the elderly, and eventually may lead to heart failure. Its surgical replacement (SAVR) was the only definitive treatment, but this operation is considered to be of increased risk for morbidity and mortality. Also, there is a growing number of elderly with severe co-morbidities, who are considered as high risk patients, that cannot undergo such an operation. Transcatheter Aortic Valve Replacement (TAVR) offered an alternative method of treatment for these patients. Furthermore, its indications were expanded to intermediate risk patients due to its advantages over SAVR.

At first, general anesthesia was the most popular anesthetic method for TAVR. However, conscious sedation and Monitored Anesthesia Care (MAC) have emerged as advantageous alternatives, in terms of inotropic drug usage, procedural times, intensive care unit (ICU) and hospital length of stay. However, few data exist about the anesthetic agents that are most suitable for TAVR under MAC, with propofol and dexmedetomidine being the most popular of them.

This is a prospective comparative study of propofol versus dexmedetomidine used for MAC in TAVR procedures. The patients will be randomly allocated into two groups and will be sedated by continuous infusion of either propofol or dexmedetomidine during the TAVR procedure. These two groups will be assessed for the overall quality of the sedation method, the clinical outcomes, the adverse events and the duration of hospitalization. At the preoperative evaluation, detailed patients' medical history will be taken, their comorbidities, physique, heart echocardiography measurements, level of frailty, renal function and neurocognitive level will be assessed and recorded and, finally, signed consent will be obtained.

During the procedure, the depth of sedation will be monitored with the use of Patient State Index (PSI) and the fluctuation of arterial pressure, heart rate, and oxygen saturation, the administration of vasoactive agents and fluids, apnea episodes and diuresis will be also recorded. By the end of the procedure, the volume and type of contrast agent used, the type of the implanted valve and the duration of both the sedation and the operation will be documented. Throughout their hospitalization, adverse events, renal function and neurocognitive level will be recorded, along with the occurrence of postoperative delirium. After patients' discharge, their duration of hospitalization, both in cardiac intensive care unit and cardiology clinic will be recorded. Follow up of the patients will be completed after thirty days. All-cause mortality will be assessed at this point and there will be a detailed recording of any adverse events and/or re-hospitalization along with long-term assessment of renal and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for TAVR

Exclusion Criteria:

* Emergency operation
* Pre-existing neurocognitive dysfunction (Mini Mental State Examination score <23)
* Inability to cooparate - communicate
* End Stage Renal Disease
* Allergy to any of the administrated drugs
* No consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Change of serum creatinine from baseline | Up to 30 days
  Assessment of renal function by serial measurements of serum creatinine (mg/dL) at four different time points (at baseline, at 24 hours, at 48 hours and at 30 days postoperatively).
Change of blood urea nitrogen (BUN) from baseline | Up to 30 days
  Assessment of renal function by serial measurements of BUN (mg/dL) at four different time points (at baseline, at 24 hours, at 48 hours and at 30 days postoperatively).
Change of serum cystatin C from baseline | Up to 30 days
  Assessment of renal function by serial measurements of serum cystatin C (mg/l) at four different time points (at baseline, at 24 hours, at 48 hours and at 30 days postoperatively).
Change of glomerular filtration rate (GFR) from baseline using the Cockcoft-Gault equation | Up to 30 days
  Assessment of renal function by serial calculations of GFR (ml/min) at four different time points (at baseline, at 24 hours, at 48 hours and at 30 days postoperatively) using the Cockcoft-Gault equation.
Change of glomerular filtration rate (GFR) from baseline using the MDRD equation | Up to 30 days
  Assessment of renal function by serial calculations of GFR (ml/min) at four different time points (at baseline, at 24 hours, at 48 hours and at 30 days postoperatively) using the MDMR equation.
Postoperative dellirium | 48 hours
  Recording of postoperative delirium using the Confusion Assessment Method (CAM) score.

SECONDARY OUTCOMES:
Death | Up to 30 days
  The occurence of death
Neurocognitive level | Up to 48 hours
  Assessment of neurocognitive function of the patient with the use of the mini mental state examination (MMSE) score.
Vasoactive and inotropic agents | Intraoperatively
  The usage of norepinephrine, epinephrine, phenylephrine, ephedrine, nitroglycerin, atropine, or other relevant agents will be recorded as the cumulative dosage of each administered during the procedure.
Stroke | Up to 30 days
  The occurrence of stroke after the procedure will be assessed as a binary outcome variable (yes/no).
Myocardial infraction | Up to 30 days
  The occurrence of myocardial infraction after the procedure will be assessed as a binary outcome variable (yes/no).
Acute heart failure | Up to 30 days
  The occurrence of acute heart failure after the procedure will be assessed as a binary outcome variable (yes/no).
Life threatening arrythmias | Up to 30 days
  The occurrence of life threatening arrythmias after the procedure will be assessed as a binary outcome variable (yes/no).
Rehospitalization | Up to 30 days
  The occurrence of rehospitalization will be assessed as a binary outcome variable (yes/no).
Pain intensity | Up to 48 hours
  Pain intensity will be recorded using the numerical rating scale (NRS).
Headache | Up to 48 hours
  The occurrence of headache after the procedure will be assessed as a binary outcome variable (yes/no)
Nausea/vomiting | Up to 48 hours
  The occurrence of nausea/vomiting after the procedure will be assessed by a 5-point scale (0 to 4, with 4 indicating the worse outcome).
Pruritus | Up to 48 hours
  The occurrence of pruritus after the procedure will be assessed by an 11-point scale (0 to 10, with 10 indicating the worse outcome).
Hypoxemia | Up to 48 hours
  The occurrence of hypoxemia after the procedure will be assessed by continuous monitoring of oxygen level (SpO2).
Duration of sedation | Intraoperatively
  The duration of sedation is defined as the time (minutes) from the start of the sedative agent administration to patient recovery (alert and able to communicate).
Procedural time | Intraoperatively
  Procedural time is defined as the time (minutes) from the start of the procedure to last suture.
Rapid pacing time | Intraoperatively
  Rapid pacing time is defined as the cumulative time (seconds) of rapid ventricular pacing performed during the procedure.
ICU length of stay | Postoperatively and up to 30 days
  The cumulative length of stay in the cardiac intensive care unit (days) after the procedure.
Length of stay | Postoperatively and up to 30 days
  The cumulative length of stay in the ward (days) after the procedure.
Patient satisfaction | 24 hours
  Patient satisfaction will be assessed using the Likert satisfaction scale.
Cardiologist satisfaction | 24 hours
  The satisfaction of the interventional cardiologists performing the procedure will be assessed by the Likert satisfaction scale.
Awareness | Up to 30 days
  Occurrence of intraoperative awareness of the patient will be assessed using the Michigan Awareness Classification Instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevas Tseniklidis, MD, Principal Investigator — University of Ioannina
Locations (1):
- Univesity Hospital of Ioannina, Ioannina, Epirus, Greece